CLINICAL TRIAL: NCT00826501
Title: Randomized Trial Comparing Endoscopy and Surgery for Pancreatic Cyst-gastrostomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shyam Varadarajulu (Other)
Responsible Party: Sponsor-Investigator, Shyam Varadarajulu, Principal Investigator, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: F080108003
Record Dates: First submitted 2009-01-20; First posted 2009-01-22 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2013-03

CONDITIONS: Pancreatic Pseudocysts
MeSH Terms: conditions — Pancreatic Pseudocyst

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Endoscopic cyst-gastrostomy with a neurolytic block along with oral/transdermal analgesic therapy
  Interventions: Procedure: Endoscopic cyst-gastrostomy
- 2 (Active Comparator): Surgical cyst-gastrostomy with neurolytic block and pain managed by only oral/transdermal analgesic
  Interventions: Procedure: Surgical cyst-gastrostomy

INTERVENTIONS:
Procedure: Endoscopic cyst-gastrostomy — After passing a small camera into the stomach the pseudocyst will be punctured and drained into the stomach by stent placement.
  Arms: 1
Procedure: Surgical cyst-gastrostomy — After making an incision in the abdomen the pseudocyst contents will be emptied and the pseudocyst will be sutured to the stomach.
  Arms: 2

SUMMARY:
Patients with pancreatitis can develop inflammatory fluid collection around the pancreas called pseudocysts. Pseudocysts may cause abdominal pain when they are more than 6cm in size. These pseudocysts can be treated (drained) by surgery or by endoscopy. Both treatment options are the current standard-of-care at all institutions around the World. The aim of this study is to identify the better of the two techniques, surgery versus endoscopy, for treatment of patients with pancreatic pseudocysts. This will be done by comparing a) the rates of pseudocyst recurrence b) quality of life of patients following treatment and c) cost associated with treatment, between both treatment modalities.

DETAILED DESCRIPTION:
The purpose of this study is to examine endoscopic ultrasound guided celiac plexus neurolysis (CPN) with analgesic therapy in patients with unresectable pancreatic cancer will decrease the severity of abdominal pain when compared to analgesic therapy alone. The specific primary aim of this study is to evaluate the efficacy of EUS-CPN + analgesic therapy (Group 1) in pain relief of patients with unresectable pancreatic cancer when compared with analgesic therapy (Group 2). The hypothesis will be tested by comparing the changes in reported pain severity between those who receive EUS-CPN in addition to analgesic therapy as compared to analgesic therapy alone.

ELIGIBILITY:
Inclusion Criteria:

* age > 19yrs
* able to provide informed consent
* pancreatic pseudocyst by CT

Exclusion Criteria:

* age < 19yrs
* unable to consent
* pancreatic abscess or necrosis

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-12 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Compare median time to pseudocyst recurrence between patients undergoing EUS or Surgical Cysto-gastrostomy | 24 months

SECONDARY OUTCOMES:
Quality of Life following treatment which will be assessed on a 3-month basis for 24-months using the SF-36 questionnaire | 24 months
Median time to pseudocyst recurrence at 24 month follow-up. | 24 months
  Median time to pseudocyst recurrence at 24 month follow-up.

OTHER OUTCOMES:
Compare pain medication usage | 24 months
  We will attempt to assess the amount of oral/transdermal opiate pain medication used in both arms to determine the efficacy of the neurolytic block.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Varadarajulu S, Bang JY, Sutton BS, Trevino JM, Christein JD, Wilcox CM. Equal efficacy of endoscopic and surgical cystogastrostomy for pancreatic pseudocyst drainage in a randomized trial. Gastroenterology. 2013 Sep;145(3):583-90.e1. doi: 10.1053/j.gastro.2013.05.046. Epub 2013 May 31. PMID 23732774